CLINICAL TRIAL: NCT01029223
Title: The Influence of Heart Rate Reduction Upon Central Arterial Pressure in Younger and Older Healthy Individuals
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Prof Bronwyn Kingwell, Baker IDI Heart & Diabetes Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 141/07
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Ivabradine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ivabradine (Experimental)
  Interventions: Drug: ivabradine
- metoprolol (Experimental)
  Interventions: Drug: metoprolol
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ivabradine
  Arms: ivabradine
Drug: metoprolol
  Arms: metoprolol
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the effect of slowing heart rate upon both central and peripheral blood pressures using a medication called Ivabradine which slows heart rate without affecting heart contraction, and to compare the effects of ivabradine to a traditional blood pressure lowering medication called metoprolol (which is a beta-blocker).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 25 years OR
* Aged > 60 years

Exclusion Criteria

* Chronic disease
* Unable to give informed consent
* Treated or untreated systemic arterial hypertension (SBP > 160 mmHg and/or DBP > 90 mmHg)
* Resting bradycardia (heart rate < 60 beats/minute)
* Pregnancy or active lactation

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
central and peripheral arterial and pulse wave velocity | baseline, and 4 hours following the administration of placebo, metoprolol or ivabradine.

SECONDARY OUTCOMES:
Central pulse pressure | Baseline measurements of central and peripheral arterial and pulse wave velocity will be made at baseline, and 4 hours following the administration of either placebo, metoprolol or ivabradine.